CLINICAL TRIAL: NCT03853642
Title: Blood Eosinophil Measurements Throughout the Day in Patients With Stable Chronic Obstructive Pulmonary Disease
Brief Title: Blood Eosinophil Measurements in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: UniversitairZB 18-409
Record Dates: First submitted 2019-02-18; First posted 2019-02-25 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-arm trial: Patient receiving blood sampling, spirometry and Feno
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling, Spirometry, Fraction exhaled Nitric Oxide
  Other Names: Spirometry and Fraction exhaled Nitric Oxide

SUMMARY:
This study will assess the within-day variation of blood eosinophils in patients with Chronic Obstructive Pulmonary disease (COPD) in stable state and determine if there is a correlation between the blood eosinophils and certain clinical parameters.

DETAILED DESCRIPTION:
COPD is a heterogeneous disease, resulting in different phenotypes with varying clinical and pathophysiological characteristics. One of these pathophysiological features is chronic airway inflammation which can be eosinophilic of nature. Blood eosinophils could be an accessible biomarker for this eosinophilic inflammation.

Eosinophil counts can fluctuate due to their short half-life in blood and due to a diurnal rhythm. More needs to be known about this diurnal rhythm and the different confounding factors and sources of within-subject variability of this biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing and able to give informed consent for participation in the study.
* Age 18 years or older.
* Diagnosis of COPD according to GOLD (Global Initiative for Chronic Obstructive Lung Disease): post-bronchodilator Tiffeneau index <0.7), in a stable state of the disease.
* A smoking history of >10 pack-years

Exclusion criteria:

* Clinical diagnosis of asthma.
* Use of systemic corticosteroids (oral, intravenous or infiltration) up to six weeks before inclusion.
* Pregnancy.
* A recent exacerbation of COPD (<4 weeks).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Within-day within-subject level changes of blood eosinophils | 12 hours
  Describe the within-day within-subject levels of blood eosinophils and determine the within-day within-subject variability of blood eosinophils

CONTACTS AND LOCATIONS:
Overall Officials: Ines Van Rossem, MD, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Universiatir Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT03853642/Prot_000.pdf